CLINICAL TRIAL: NCT02579902
Title: Effect of Vitamin D3 Supplementation on Clinical Signs, Oxidative Stress and Inflammatory Biomarkers in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Vitamin D3 Supplementation in Treatment of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Abbasnezhad, Ph.D candidate of Nutrition Sciences, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ir.ajums.rec.1394.306
Record Dates: First submitted 2015-10-11; First posted 2015-10-20 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; inflammation; oxidative stress; clinical signs; vitamin D3
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation; Signs and Symptoms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vitamin D3 (Active Comparator): 50000 IU vitamin D3 capsule, one capsule every 2 weeks for 6 months.
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)
- placebo (Placebo Comparator): Placebo capsule, one capsule every 2 weeks for 6 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (Cholecalciferol) — 50000 IU Vitamin D3 (Cholecalciferol) will be given as one gelcaps every 2 weeks for a period of 6 months.
  Arms: Vitamin D3
Dietary Supplement: placebo — placebo will be given in identical gelcaps once every 2 weeks for a period of 6 months.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether vitamin D3 supplementation is effective in the treatment of clinical signs, biomarkers of inflammation and oxidative stress due to Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
This randomized double blind clinical trial will be performed on 90 patients (45 in intervention and 45 in control group) diagnosed with IBS. The intervention group will receive 50000 IU vitamin D3 and the control group will receive placebo contains edible paraffin once every 2 weeks for six months. Variables including biomarkers of inflammation and oxidative stress, serum levels of calcium and vitamin D, anthropometric indicators and blood pressure will be measured at baseline and end of the study. The investigators will use Rome III questionnaire for evaluating the clinical signs of the disease. The questionnaires will be filled out at baseline and every 2 weeks by the patients for six months.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are diagnosed with Irritable Bowel Syndrome (IBS) according to ROME III criteria; Signed consent by the patient.

Exclusion Criteria:

* Patients who have celiac disease (diagnosed by a duodenal biopsy or celiac serological tests)
* Any other diseases of the gastrointestinal tract such as Inflammatory Bowel Disease (IBD)
* Any kind of abdominal surgery
* Chronic disease such as diabetes
* Cardiovascular, hepatic
* Kidney and severe infection
* Pregnancy
* Breastfeeding
* Smoking
* Alcohol consumption
* Use of dietary supplements
* Use of vitamin D and calcium supplement during the last year before the study
* Use any medication for signs improvement during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical signs including abdominal pain, bloating, rumbling, abdominal distention, dissatisfaction with stool consistency | up to six months
  clinical signs will be assessed by Visual Analog Scale (VAS) 0-100mm self-report questionnaire at baseline and every two weeks for six months.
Symptom Severity Score | up to six months
  symptom severity score will be assessed by IBS-Symptom Severity Score (IBS-SSS) self-report questionnaire baseline and after six months intervention.

SECONDARY OUTCOMES:
Dietary intake | up to six months
  24-Hour dietary recalls questionnaires will be used to assess dietary pattern at baseline and after 3 and 6 months intervention.
Body Weight | up to six months
  Body Weight will be measured in kilograms at baseline and after six months intervention.
Body Mass Index (BMI) | up to six months
  BMI is weight in kilograms divided to height in meters squared. It will be measured at baseline and after six months intervention.
Waist Circumference (WC) | up to six months
  WC will be measured in centimeter at baseline and after six months intervention.
Hip Circumference (HC) | up to six months
  HC will be measured in centimeter at baseline and after six months intervention.
Waist to Hip Ratio (WHR) | up to six months
  WHR is WC divided to HC. It will be measured at baseline and after six months intervention.
Blood Pressure (BP) | up to six months
  BP will be measured in mmHg at baseline and after six months intervention.
Health-related Quality of Life | up to six months
  Health-Related Quality of Life will be assessed by IBS-Quality Of Life (IBS-QOL) with 34-item Short-Form (SF-34) self-report questionnaire at baseline and after six months intervention.
Tumor Necrosis Factor-α (TNF-α) | up to six months
  Blood serum TNF-α will be assessed by enzyme-linked immunosorbent assay (ELISA) at baseline and after six months intervention.
Interleukin-10 (IL-10) | up to six months
  Blood serum IL-10 will be assessed by ELISA at baseline and after six months intervention.
Interleukin-17 (IL-17) | up to six months
  Blood serum IL-17 will be assessed by ELISA at baseline and after six months intervention.
Malondialdehyde (MDA) | up to six months
  Blood serum MDA will be assessed by Thiobarbituric acid (TBA) method at baseline and after six months intervention.
Total Antioxidant Capacity (TAC) | up to six months
  Blood serum TAC will be assessed by Ferric Reducing Antioxidant Power (FRAP) assay at baseline and after six months intervention.
25-hydroxy vitamin D (25(OH)D) | up to six months
  Blood serum 25(OH)D will be assessed by Radioimmunoassay at baseline and after six months intervention.
Calcium | up to six months
  Blood serum Calcium will be assessed by Arsenazo III method at baseline and after six months intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Ahvaz Jundishapur University of Medical Sciences, Ahvāz, Khuzestan, Iran